CLINICAL TRIAL: NCT05666778
Title: Single Arm Trial of Menstrual Cups Among Economically Vulnerable Women to Reduce Bacterial Vaginosis and STIs Through Reduced Harmful Sexual and Menstrual Practices
Brief Title: Single Arm Trial of Menstrual Cups Among Economically Vulnerable Women to Reduce Bacterial Vaginosis and STIs
Acronym: POWWERHealth
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Nyanza Reproductive Health Society (Other); Liverpool School of Tropical Medicine (Other); University of Illinois at Chicago (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 22040505; R01AI170564 (NIH)
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Bacterial Vaginosis; Vaginal Microbiome; Chlamydia Trachomatis Infection; Neisseria Gonorrheae Infection; Trichomonas Vaginitis
Keywords: Menstrual Cup; Menstrual Health; Menstrual Hygiene; Bacterial vaginosis; Vaginal microbiome; Sexually transmitted infections; Kenya
MeSH Terms: conditions — Vaginosis, Bacterial; Gonorrhea; Trichomonas Vaginitis; Sexually Transmitted Diseases | interventions — Menstrual Hygiene Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Other): After completing 12 months observation of usual practices of menstrual hygiene management, all participants will be provided reusable menstrual cups that can be worn during sex. The menstrual cup training is comprised of a 2 hour group session that covers basic information on reproductive health, menstrual health, and menstrual hygiene, cup use (insertion/removal), storage, cleaning. In the first three months after intervention delivery, there are monthly phone calls to assess usage and for trouble shooting. There are 12 months of observation in the menstrual cup arm, with Bacterial vaginosis (BV) and vaginal microbiome (VMB) assessment at the beginning of the 12-month period, at 6 months, and at 12 months. Sexually transmitted infection (STI) is measured at the beginning of the 12- month intervention period, and then at 12 months.
  Dec 2025: As a supplemental analysis, observation of the menstrual cup arm is extended to 18-24 months, to more fully capture putative secular trends.
  Interventions: Device: Menstrual Cup

INTERVENTIONS:
Device: Menstrual Cup — Menstrual cups are inserted vaginally to collect menstrual flow, with some designed especially for use during intercourse, which will be used in this study. Medical devices registered with the U.S. FDA, a reusable silicon cup can last up to 10 years, is cost-effective, and has reduced environmental impact.

SUMMARY:
HIV remains a global pandemic with 37 million infected. In western Kenya, 16% of women in the general population and 29% of the poorest women have HIV. The HIV and sexually transmitted infection (STI) epidemics overlap with broader reproductive health concerns. Menstrual hygiene management is a big problem in low- and middle-income countries and a lack of menstrual products negatively impacts women's work-life. This comes from cultural taboos, stigma, and discrimination, promoting secrecy around menstruation, high cost of menstrual products, use of traditional materials (e.g. rags, cotton wool, etc.) causing leakage and odor, and lack of water and safe hygiene facilities. Menstrual cups designed for use during sex may help women prevent Bacterial vaginosis (BV) and STIs through hygienic period practices, and may help them avoid bad practices in an attempt to maintain vaginal dryness. The goal of this interventional trial is to test the impact of menstrual cups on vaginal microbiome, BV, and STIs of poor women at high risk for STIs and HIV. We predict to see 25% less BV, our primary outcome, over one year. This trial aims to learn more about the safety of the intervention, and understand what is needed to fully implement the program.

DETAILED DESCRIPTION:
In western Kenya, HIV prevalence is 16% among women in the general population, and 29% among the most economically constrained women. The HIV/STI epidemic overlaps with broader reproductive health concerns. Menstrual hygiene management (MHM) is a pervasive problem across low- and middle-income countries. In Phillips-Howards' survey of over 3,400 women in rural Kenya, two-thirds of women in impoverished settings state they depend on their sexual partners to provide branded products. Economically vulnerable women at high risk for HIV and STI are uniquely challenged because many continue to have sex during menses, and engage in harmful MHM practices, such as vaginal insertion of sponges and cotton to maintain dryness. Led by co-investigator Phillips-Howard, a cluster-randomized study of 644 girls aged 14-16 years old in western Kenya compared reusable menstrual cups to usual menstrual practice and counseling; after 9 months, menstrual cup use resulted in 35% reduction (p=0.034) in Bacterial vaginosis (BV) prevalence and 56% reduction (p=0.001) in STI prevalence compared to other materials. Among 431 Kenyan secondary schoolgirls aged 14-21, we observed cloth use for menses was associated with a 1.72-fold increased odds of non-optimal vaginal microbiome (CST-IV vs. CST-I: aOR=1.90; 95% CI: 1.03-2.86). Over 18 months of observation prior to COVID-19, girls using menstrual cups to manage menses had 20% higher occurrence of Lactobacillus crispatus dominated CST-I (aRR=1.29; 95% CI: 1.08-1.53, controlling for age, and baseline STI and sexual activity). Menstrual cups designed for use during intercourse may help women prevent BV and STIs through hygienic menstrual practices and avoidance of harmful practices to maintain vaginal dryness during menses. Objective: This single-arm interventional trial seeks to evaluate the preliminary efficacy of menstrual cups on non-optimal vaginal microbiome (VMB), BV, and STIs of economically vulnerable women at high risk for STIs and HIV, assess safety profile, and understand implementation needs. In Aim 1, we will evaluate the impact of menstrual cups on VMB, BV, and STIs among 402 economically vulnerable women in semi-urban Kenya. In Aim 2, we will conduct integrated surveillance for enhanced detection of safety endpoints, risk of cup contamination, and mitigating or facilitating water, sanitation, hygiene (WASH) factors. In Aim 3, we will identify constructs for successful MHM program implementation using an implementation science framework. Future Directions: The biological protection suggested in a randomized setting, and our findings that unhygienic cloth use is associated with non-optimal VMB, while menstrual cup use increases optimal VMB composition, together provide rational justification for this trial, of relevance to economically challenged women globally. Assessing preliminary efficacy signal in conjunction with implementation characteristics and adverse events, will generate a comprehensive and necessary foundation for definitive assessment of effectiveness of menstrual cups as a multipurpose intervention for MHM, and to reduce BV and STIs.

ELIGIBILITY:
Inclusion Criteria:

* age 15-35 years,
* able to provide informed consent,
* residing in Kisumu County,
* not currently pregnant,
* has experienced a menstrual period in the past 2 months, and
* dependent on sex for livelihood as defined above.

Exclusion Criteria:

* pregnancy,
* post-natal (within 6 months),
* post-menopausal,
* amenorrhea,
* IUD in situ.

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — The interventional portion of this study includes only cis-gendered females, as outcomes related to the vaginal microbiome and menstruation are relevant only to biological females. To illustrate how menstrual hygiene management may biologically mediate the vaginal microbiome and subsequent related outcomes of BV and STIs, it is essential to enroll females.
Enrollment: 408 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of menstrual cups on BV | 2 years
  For primary outcome BV (binary, 7-10 vs. 0-6) the measures will be baseline to 12 month cumulative incidence control/pre-menstrual cup intervention and 12- to 24-month cumulative incidence in the intervention phase. We will employ a linear mixed model (LMM; observations nested in individual), with binomial distribution and log link function, examining cup use as a time-varying exposure among all participants who were given the cup within the intervention phase and reported using the cup. A supplemental analysis may examine BV from 12-36 months in the intervention phase.

SECONDARY OUTCOMES:
Evaluate the impact of menstrual cups on STI | 2 years
  We employ similar approach for analysis of secondary outcome of STI (binary composite of infection with Chlamydia trachomatis [CT], Neisseria gonorrhoeae [NG], or Trichomonas vaginalis [TV]), as for Outcome 1.
Evaluate the impact of menstrual cups on vaginal microbiome (VMB) | 2 years
  Vaginal microbiome will be dichotomized as Community State Type I (CST-I; Lactobacillus crispatus dominated; optimal) vs. other CST. We will employ similar approach for analysis of secondary outcome of VMB (binary) as for Outcome 1.

CONTACTS AND LOCATIONS:
Locations (2):
- Rush University Medical Center, Chicago, Illinois, United States
- Nyanza Reproductive Health Society, Kisumu, Nyanza, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Minimum IPD for main analysis replication will be made available at the time of publication. After completion of the study, data will be deposited in a registry for clinical trials data within 15 months.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: ICFs and analytic code, will be included as supplementary material with published with manuscripts.

REFERENCES:
- [Derived] Zulaika G, Otieno FO, Mason L, van Eijk AM, Bhaumik R, Green SJ, Phillips-Howard PA, Mehta SD. Menstrual cups to reduce bacterial vaginosis and STIs through reduced harmful sexual and menstrual practices among economically vulnerable women: protocol of a single arm trial in western Kenya. BMC Public Health. 2024 Nov 8;24(1):3089. doi: 10.1186/s12889-024-20491-z. PMID 39516733